CLINICAL TRIAL: NCT06751537
Title: Effectiveness of WearME System for FEV1/FVC, Respiration and Activity Biomarkers in COPD Patients
Brief Title: Effectiveness of the WearME System for COPD Severity and Respiratory Function
Acronym: WearME-COPD
Status: Recruiting | Type: Observational
Sponsor: LASARRUS Clinic and Research Center (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University (Other); Tidalhealth (Unknown); Tidalhealth, Inc. (Unknown); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Other Study IDs: LAS-01-WZ-023; 1R44HL172444-01A1 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: lung function; respiratory rate; FEV1; FVC; I:E ratio; Pulmonary Devices; Machine Learning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD Participants: Participants are wearing the WearME device and undergoing reference testing

SUMMARY:
This observational study evaluates the effectiveness of the WearME system in monitoring COPD severity and respiratory function by comparing its measurements to standard spirometry, capnography, and other clinical assessments in 128 COPD participants.

DETAILED DESCRIPTION:
COPD is the third leading cause of death worldwide, with over 3 million deaths and an estimated total cost of $52 billion in the U.S. alone. This project, in collaboration with the Johns Hopkins Clinical Research Network (JHCRN), aims to provide technological innovation access to underserved patients in low-income, rural, and diverse ethnicities in the Mid-Atlantic region.

The symptoms of COPD include dyspnea (shortness of breath), coughing and the production of sputum. Recent data shows that the 30-day readmission rate of COPD patients is approaching 23%, creating a huge burden on the health care system. Exacerbations can commonly be treated in the home if detected early, so early recognition of symptoms signaling an impending COPD exacerbation may reduce readmission and associated healthcare costs. The standard adjuncts used to assess lung function (e.g., spirometry, plethysmography, CT scan) require oversight by medical experts, are time consuming, and do not allow for continuous and remote patient monitoring of an acute exacerbation. Early recognition of deteriorating patient's lung function will enable timely intervention and help manage changes in COPD severity.

2. EFFECTIVENESS STUDY OVERVIEW

In this study, the WearME-Basic functionality will be validated while using the same hardware needed for the WearME-Basic app. Since the hardware collects all data needed to supply either the Basic or Pro app, the investigators will also gain insights on both the Basic and Pro simultaneously during this study.

This study will assess the effectiveness of the WearME-Pro system in monitoring COPD patients by measuring the accuracy and reliability of the system for forced expiratory volume (FEV₁), forced vital capacity (FVC), respiratory rate, heart rate, I:E ratio, spinal range of motion (ROM), and activity levels. Up to 128 COPD participants will be recruited from the LASARRUS outpatient clinic, Johns Hopkins and TidalHealth hospitals, and stratified into four groups based on the GOLD standard for severity stratification. Participants will be asked to wear the WearME system during a data collection period of 145 minutes.

The primary outcome measure will be the Bland-Altman LOA between the FEV1/FVC measurements of WearME-Pro FEV1/FVC prediction (recorded within the WearME-Basic app but not displayed to users) and the gold standard devices. Secondary outcomes include the validation of the WearME-Basic system for FDA submission by evaluating its accuracy in measuring respiration rate, heart rate, I:E ratio, and ROM compared to gold standard reference devices, and correlation of I:E measured by the WearME device to FEV1/FVC measured by spirometry.

We will use standard medical devices as reference devices for comparison with the WearME systems outputs. The specific devices used for spirometry, capnography, heart rate monitoring, and range of motion measurement will be appropriate, FDA-cleared devices commonly used in clinical practice.

Details of the specific device models and their usage will be documented in the Manual of Procedures (MOP). The sponsor will provide all necessary reference devices to the study sites, including the spirometers, capnographs, and other equipment required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants aged 21-100 years, of any sex, and of any race/ethnicity, who are able to understand and sign consent documents in English or Spanish.
* Diagnosed with COPD as per the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria [5] , with the following severity levels (confirmed via spirometry performed after consent):

  * Mild: FEV1/FVC < 0.7 and FEV1 ≥ 80%
  * Moderate: FEV1/FVC < 0.7 and 50% ≤ FEV1 < 80%
  * Severe: FEV1/FVC < 0.7 and 30% ≤ FEV1 < 50%
  * Very Severe: FEV1/FVC < 0.7 and FEV1 < 30% or FEV1 < 50%, plus chronic respiratory failure.

Note: Participants will be consented and enrolled based on prior diagnosis of COPD from medical records within the past year to confirm eligibility and stratify COPD severity levels. Spirometry will be performed during concurrent data collection with the WearME device for comparison. Screening failures are expected and will be recorded and managed appropriately.

* Current, former, or never smoker; any amount of time between quitting and study enrollment is allowed).
* Ability to understand and willingness to sign consent documents.
* Able to participate in study procedures as required.

Exclusion Criteria:

* Participants with known skin allergies or conditions that may interfere with device application or signal transmission.
* Currently receiving invasive mechanical ventilation.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult COPD patients recruited from outpatient clinics at LASARRUS, Johns Hopkins, and TidalHealth.
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Agreement between WearME-Pro system and gold standard devices for FEV1 measurements, stratified by COPD severity. | Within 6 months of study start.
  The primary outcome measure will be the Bland-Altman LOA between the FEV1/FVC measurements of WearME-Pro FEV1/FVC prediction (recorded within the WearME-Basic app but not displayed to users) and the gold standard devices.

SECONDARY OUTCOMES:
Accuracy of WearME-Basic in measuring Respiration Rate | Within 6 months of study start.
  Accuracy of WearME-Basic in measuring Respiration Rate
Accuracy of WearME-Basic in measuring I:E ratio | Within 6 months of study start.
  Accuracy of WearME-Basic in measuring I:E ratio
Accuracy of WearME-Basic in measuring Heart Rate | Within 6 months of study start.
  Accuracy of WearME-Basic in measuring Heart Rate
Accuracy of WearME-Basic in measuring ROM | Within 6 months of study start.
  Accuracy of WearME-Basic in measuring ROM

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins, Baltimore, Maryland
  - TidalHealth, Salisbury, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Data Types:
  Scientific Data to be Shared:
  1. Clinical Data:
     * De-identified patient demographics (age, sex, ethnicity)
     * Clinical assessments and outcomes
     * Pulmonary function test results (e.g., FEV1, FVC ratios)
     * Respiratory rate (RR), Inspiratory/Expiratory (I:E) ratio, activity measurements
  2. Physiological Measurements:
     * Bilateral acoustic recordings from the WearME-Pro device
     * Kinematic data (accelerometer, gyroscope readings)
     * Temperature measurements
  3. Machine Learning Outputs:
     * Model parameters and outputs from the AUDAS algorithm
     * Processed data used for developing predictive models
  Data Sharing and Access:
  1. Repository Selection: Upon completion of the project, de-identified datasets and associated metadata will be deposited in Figshare, a widely used, NIH-compliant public repository that provides persistent identifiers (DOIs) and facilitates open access.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Nicholson PJ. The updated ATS/ERS spirometry technical standards. Occup Med (Lond). 2020 May 27;70(3):146-148. doi: 10.1093/occmed/kqaa030. No abstract available. PMID 32073625
- [Background] Lokke A, Lange P, Lykkegaard J, Ibsen R, Andersson M, de Fine Licht S, Hilberg O. Economic Burden of COPD by Disease Severity - A Nationwide Cohort Study in Denmark. Int J Chron Obstruct Pulmon Dis. 2021 Mar 10;16:603-613. doi: 10.2147/COPD.S295388. eCollection 2021. PMID 33731990
- [Background] GBD Chronic Respiratory Disease Collaborators. Prevalence and attributable health burden of chronic respiratory diseases, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Respir Med. 2020 Jun;8(6):585-596. doi: 10.1016/S2213-2600(20)30105-3. PMID 32526187